CLINICAL TRIAL: NCT03757325
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL747 in Subjects With Alzheimer's Disease
Brief Title: Study to Evaluate DNL747 in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-D-0002
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DNL747 First, Placebo Second (Experimental): Subjects will receive DNL747 for 29 days for the first period and then will switch to placebo for 29 days for the second period. There will be a 14-day washout period between the 2 treatment periods.
  Interventions: Drug: DNL747; Drug: Placebo
- Placebo First, DNL747 Second (Experimental): Subjects will receive placebo for 29 days for the first period and then will switch to DNL747 for 29 days for the second period. There will be a 14-day washout period between the 2 treatment periods.
  Interventions: Drug: DNL747; Drug: Placebo

INTERVENTIONS:
Drug: DNL747 — DNL747
Drug: Placebo — Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple oral doses of DNL747 in subjects with Alzheimer's disease when administered for 29 days in a cross-over design

DETAILED DESCRIPTION:
This is a Phase 1b randomized, placebo-controlled, double-blind, crossover study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of DNL747 in subjects with Alzheimer's disease (AD)

ELIGIBILITY:
Key Inclusion Criteria:

* Women of non-childbearing potential and men, aged 55-85 years
* AD diagnosis based on the 2011 National Institute on Aging-Alzheimer's Association Guidelines
* Supportive evidence for diagnosis of AD based upon positive CSF Aβ42 test, or documented history of positive amyloid-specific PET scan
* Screening MMSE score of 16-26 points
* Screening CDR Global Score of 0.5-1.0
* Availability of a person ("caregiver") who, in the investigator's judgment, has frequent and sufficient contact with the participant and is able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to provide information at clinic visits that require input for scale completion, assists the participant with compliance for at-home study treatment administration, and signs the necessary consent form (note: the caregiver is not required to stay in the unit)
* Approved AD treatments (acetylcholinesterase inhibitors ± memantine) and other prescription medications must be stable for ≥1 month prior to screening and anticipated to be stable over the duration of the study

Key Exclusion Criteria:

* Clinical history within 2 years of the screening visit or current evidence of any neurological or neurodegenerative disorder other than AD that is associated with transient or sustained alterations in cognition
* Magnetic resonance imaging (MRI) at screening (or within 1 year of screening visit) consistent with any neurological or neurodegenerative disorder other than AD that is associated with transient or sustained alterations in cognition

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Randomization - Day 86
Number of Subjects with clinically significant neurological examination abnormalities | Randomization - Day 86
Number of Subjects with laboratory test abnormalities | Randomization - Day 86

SECONDARY OUTCOMES:
Pharmacokinetic measure of maximum observed plasma concentration (Cmax) of DNL747 | Randomization - Day 86
Pharmacokinetic measure of time to reach maximum observed plasma concentration (Tmax) of DNL747 | Randomization - Day 86
Pharmacokinetic measure of area under the plasma drug concentration-time curve (AUC) of DNL747 | Randomization - Day 86
Pharmacokinetic terminal disposition rate constant (λz) with the respective t1/2 of DNL747 | Randomization - Day 86
Pharmacokinetic measure of CSF concentrations of DNL747 | Randomization - Day 86
Pharmacodynamic measure of pS166 in PBMCs | Randomization - Day 86

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Clinical Site(s), Miami, Florida
  - Clinical Site(s), Orlando, Florida
  - Clinical Site(s), Dallas, Texas
  - Clinical Site(s), Salt Lake City, Utah
- Clinical Site(s), Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vissers MFJM, Heuberger JAAC, Groeneveld GJ, Oude Nijhuis J, De Deyn PP, Hadi S, Harris J, Tsai RM, Cruz-Herranz A, Huang F, Tong V, Erickson R, Zhu Y, Scearce-Levie K, Hsiao-Nakamoto J, Tang X, Chang M, Fox BM, Estrada AA, Pomponio RJ, Alonso-Alonso M, Zilberstein M, Atassi N, Troyer MD, Ho C. Safety, pharmacokinetics and target engagement of novel RIPK1 inhibitor SAR443060 (DNL747) for neurodegenerative disorders: Randomized, placebo-controlled, double-blind phase I/Ib studies in healthy subjects and patients. Clin Transl Sci. 2022 Aug;15(8):2010-2023. doi: 10.1111/cts.13317. Epub 2022 Jun 1. PMID 35649245